CLINICAL TRIAL: NCT07311044
Title: Cardiovascular Disease/ Pulmonary Hypertension and Voice Characteristics Study
Brief Title: CVD/PH and Voice Characteristics
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Other Study IDs: 20-011269
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension, Pulmonary; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the association between patient voice signal characteristics and the presence and severity of pulmonary hypertension in patients referred for elective clinically indicated echocardiography for at Mayo Clinic MN.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who present for a routine elective, clinically indicated, diagnostic echocardiogram at the echocardiography laboratory at Mayo Clinic
* All individuals who have had a clinically indicated, diagnostic echocardiogram at the echocardiography lab at Mayo Clinic before a scheduled procedure in the cardiac catheterization lab at Mayo Clinic
* All individuals who have had a clinically indicated diagnostic echocardiogram at the echocardiography lab at Mayo Clinic and have an appointment in any CV outpatient clinic.

Exclusion Criteria:

* Known history of voice disorder either primary or secondary to neuromuscular or other pathology
* Patients under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from a list of patients scheduled for a clinically indicated echocardiogram.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of confirmed pulmonary hypertension diagnoses based on voice recording analysis | Baseline
  A successful diagnosis of pulmonary hypertension will be confirmed by echocardiogram.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No